CLINICAL TRIAL: NCT02451540
Title: Placebo Controlled Study to Assess the Effect of Roflumilast in Hyperinflated COPD Patients in Addition to LABA/LAMA Therapy Using Functional Respiratory Imaging.
Brief Title: Evaluation of the Effect of Roflumilast in Hyperinflated COPD Patients Using Functional Respiratory Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No new investigational product can be delivered to the site.
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLUI-2014-134
Record Dates: First submitted 2015-05-07; First posted 2015-05-22 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; dynamics hyperinflation; Computed Tomography scan; CT scan; Functional Respiratory Imaging; FRI; Roflumilast; PRO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator): Patient will take Roflumilast (500 micrograms) once a day for 3 months. A HRCT scan will be taken at baseline and after 3 months of treatment
  Interventions: Radiation: HRCT scan; Drug: Roflumilast
- Placebo (Placebo Comparator): Patient will take the Placebo of Roflumilast once a day for 3 months. A HRCT scan will be taken at baseline and after 3 months.
  Interventions: Radiation: HRCT scan; Drug: Placebo of Roflumilast

INTERVENTIONS:
Radiation: HRCT scan — HRCT scan of thorax, at baseline and after 3 months
Drug: Placebo of Roflumilast — Placebo, once a day in the morning during 3 months
  Other Names: Placebo
  Arms: Placebo
Drug: Roflumilast — Roflumilast, once a day in the morning during 3 months
  Other Names: Daxas
  Arms: Roflumilast

SUMMARY:
In this study the efficacy of Roflumilast in addition to LAMA/LABA therapy will be assessed using Functional Respiratory Imaging.

In total 40 Chronic obstructive pulmonary disease (COPD) patients, Global Initiative for Chronic Obstructive Lung Disease (GOLD) stages C and D, who are stable on LABA/LAMA therapy and who are prone to dynamics hyperinflation will be included in this study. To indicate the susceptibility to dynamics hyperinflation patients should have a baseline Borg Fatigue score after the 6-minute walk test (6MWT) above 4.

The patients will be randomized in such a way that 1 out of 2 patients will receive placebo and 1 the active component.

Image parameters will be assessed and the correlation with lung function and health related quality of life will be checked before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 30 years old
* Written informed consent obtained
* Patient with Body mass index (BMI) ≥ 20
* Female patient of childbearing potential who confirm that a contraception method was used at least 14 days before visit 1 and will continue to use a contraception method during the study
* COPD patient with GOLD stages C and D
* Patient with a Borg Fatigue score after the 6MWT on screening above 4 to indicate the susceptibility to dynamics hyperinflation
* Patient with smoking history of at least 10 pack-years
* Patient takes a combination therapy of LABA/ LAMA at least 6 weeks before visit 1
* Patient must be able to understand and complete the protocol requirements, instructions, questionnaires and protocol-stated restrictions

Exclusion Criteria:

* Pregnant or lactating females
* Patient with severe immunological diseases and/ or severe acute infectious diseases
* Patient with heart failure as documented in the medical history or as defined by the investigator during the physical examination performed at visit 1
* Patient with diagnosis of cancer (except basal cell carcinoma)
* Patient with a history of depression associated with suicidal ideation or behaviour
* Patient with moderate or severe hepatic impairment.
* Patient with lactose intolerance
* Patient is unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
* Patient who received inhalation corticosteroids (ICS) within the last 6 weeks prior to the screening visit
* Patient who received any investigational new drug within the last 4 weeks prior to the screening visit or twice the duration of the biological effect of any drug (whichever is longer)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in Airway volume (iVaw) | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Changes in Airway resistance (iRaw) | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Changes in Lobe volumes (iVlobes) | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Changes in Air trapping | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Changes in Internal Lobar Airflow Distribution | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Low Attenuation or Emphysema Score | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Changes in Blood Vessel Density | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Changes in Airway Wall Thickness | 3 months
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.
Aerosol deposition concentrations | At baseline and after 3 months of treatment
  By using Functional Respiratory Imaging the efficacy of Roflumilast in addition to long-acting muscarinic antagonist (LAMA)/ long acting β2-agonist (LABA) therapy will be assessed.

SECONDARY OUTCOMES:
Changes in Spirometry | At baseline and after 3 months of treatment
  Spirometry is a composite outcome measure consisting of the following parameters:
  * FEV1
  * Peak Expiratory Flow (PEF)
  * Forced Vital Capacity (FVC)
  * Maximum Expiratory Flow at 50% of FVC (MEF 50)
  * Maximum Expiratory Flow at 25% of FVC (MEF 25)
Changes in Body plethysmography | At baseline and after 3 months of treatment
  Body plethysmography is a composite outcome measure consisting of the following parameters:
  * Residual Volume (RV)
  * TLC
  * FRC
  * Airway resistance (Raw)
Changes in Diffusion capacity | At baseline and after 3 months of treatment
  Diffusion capacity is a composite outcome measure consisting of the following parameters:
  * carbon monoxide transfer factor (TCO)
  * Alveolar volume (VA)
Changes in 6MWT | At baseline and after 3 months of treatment
  Exercise capacity: distance walked in 6 minutes (m), oxygen saturation measurement will be performed during the test
Changes in Patient Related Outcome (PRO) | At baseline and after 3 months of treatment
  Patient Related Outcome is a composite outcome measure consisting of the following questionnaires:
  * Borg CR10 Scale: measure of the present dyspnea and leg fatigue before and after exercise
  * COPD assessment test (CAT): measure of the impact of COPD on your life
  * Saint George's Respiratory Questionnaire (SGRQ): measure health related quality of life and comfort

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, M.D., M.S., Principal Investigator — University Hospital of Antwerp
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerp, Belgium